CLINICAL TRIAL: NCT07165600
Title: Yoga to Improve Disparities in Cancer Survivorship
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25802; NCI-2025-05225 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Survivorship; Cancer
Keywords: Cultural support services
MeSH Terms: conditions — Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Yoga Intervention (Experimental): Participants receive a 4-week yoga intervention consisting of weekly 60-minute yoga sessions led by a trained facilitator. Participants may also participate remotely. At the end of the program, participants will also receive access to online yoga training videos (created by the study team) to continue self-practice.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Physical activity
  Other Names: Yoga training; Yoga sessions

SUMMARY:
This clinical trial tests the impact of a racially concordant trainer led yoga program on quality of life and symptom burden in Black and/or African American cancer survivors. Black individuals in the United States are more affected by cancer, despite modern advances. Cancer treatments can impact physical and mental health and overall quality of life and Black individuals report worse physical function and quality of life and less access to culturally appropriate support services. Yoga has been shown to have a positive impact on cancer and cancer treatment related symptoms and quality of life, however, a one size fits all approach has not been shown to be effective in diverse populations. A trainer that shares the same racial or ethnic background as the participant (racially concordant) may have a positive impact on communication, trust, and may improve accessibility and participation. Participating in a yoga program led by a racially concordant trainer may improve quality of life and symptom burden in Black and/or African American cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility and acceptability of a yoga intervention among Black individuals with cancer.

SECONDARY OBJECTIVES:

I. To estimate the effect of the intervention on health-related quality of life.

II. To estimate the effect of the intervention on symptom burden. III. To determine the safety of the intervention.

OUTLINE:

Participants engage in racially concordant trainer led yoga sessions over 60 minutes once weekly (QW) on weeks 1-4 then participate in self-practice video led yoga sessions over 10-15 minutes on weeks 5-8.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years.
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
4. Diagnosed with any malignancy and/or received any cancer directed therapy within 5 years of enrollment.
5. Be able to speak, read and write in English.
6. Self-identify as Black or African American race.
7. Reside in California.

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.

   a. Participants complete the PAR-Q at screening to ensure that they are physically well enough to enroll in the study. If they report any conditions that may be contraindications to physical activity, physician clearance will be required prior to enrollment.
2. Planned major surgery during the study period.
3. Any major injuries that limit physical activity.
4. Plans to receive any form of further cancer therapy during the study period (exception: individuals with breast or prostate cancer are allowed to be on hormone therapy on the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall completion rate | Up to 8 weeks
  The completion rate is defined as the proportion of enrolled individuals who attend at least 2 yoga sessions.
Median score on the Feasibility of Intervention Measure (FIM) | Up to 8 weeks
  The FIM is a four-item measure of implementation that assesses participants perceived appropriateness of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4.
Median score on the Acceptability of Intervention Measure (AIM) | Up to 8 weeks
  The AIM is a four-item measure of implementation that assesses participants perceived acceptability of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4.
Median score on the Intervention Appropriateness Measure (IAM) | Up to 8 weeks
  The IAM is a four-item measure of implementation that assesses participants perceived appropriateness of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4.

SECONDARY OUTCOMES:
Change in scores on the Patient Reported Outcomes Measurement Information System (PROMIS®-29) (Version 2) score | Up to 8 weeks
  The PROMIS 29 v2.0 profile assesses pain intensity using a response scale for each item ranging from 0 (no pain) to 10 (worst imaginable pain) on seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance), with four items per domain and one question which addresses pain intensity item. PROMIS-29 domains are scored using a T-score metric, with higher scores indicate higher levels of functioning.
Percentage of participants reporting adverse events | Up to 8 weeks
  The effect of the intervention on symptom burden will be evaluated by participants self-reporting of adverse events. Adverse events will be classified and graded according to the Common Terminology Criteria for Adverse Events (CTCAEv 5).

CONTACTS AND LOCATIONS:
Overall Officials: Sorbarikor Piawah, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No